CLINICAL TRIAL: NCT00287638
Title: To Assess the Differences in Chemokines and Oxidative Stress Markers in Exhaled Breath Condensate of Obstructive Sleep Apnoea Patients
Brief Title: Markers in Exhaled Breath Condensate in Obstructive Sleep Apnoea (OSA) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Fanny WS Ko, The Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Resp/ko/2006/002
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

ARMS (2):
- 1 (Active Comparator): CPAP
  Interventions: Device: CPAP
- 2 (Placebo Comparator): no CPAP
  Interventions: Device: placebo

INTERVENTIONS:
Device: CPAP — Continuous positive pressure device with a time clock
  Arms: 1
Device: placebo — no CPAP
  Arms: 2

SUMMARY:
Patients with obstructive sleep apnoea (OSA) have repetitive episodes of partial or complete upper airway obstruction during sleep. This leads to sleep fragmentation and symptoms like excessive daytime sleepiness and impaired psychosocial well-being. More evidence now suggested OSA is associated with cardiovascular diseases like hypertension, myocardial infarction, pulmonary hypertension and stroke.

The upper airway structure and function are altered in OSA. Some studies suggested that an increase in the levels of systemic biomarkers of inflammation and oxidative stress in patients with OSA. So far, there is only very limited data on non-invasive monitoring of inflammation involved in the upper airway of OSA patients. The inflammatory mechanisms involved in the upper airway may give some insights to the systemic effect, like cardiovascular complications, of OSA.

Measurement of the constituents of exhaled breath and exhaled breath condensate (EBC) is a non-invasive method to assess the degree of inflammation of the airway. Exhaled nitric oxide (eNO) can be measured with the subject exhaling to a mouthpiece connected to a machine measuring real-time eNO level. With the subject exhaling to a cooling unit, EBC can be collected as liquid is formed as a result of condensation.

This study will assess the eNO in exhaled breath, oxidative stress marker (8-isoprostane) and cellular inflammatory markers (eotaxin, monocyted derived chemokine, growth related oncogene- alpha, monocyte chemoattractant protein-1) in the EBC and blood of OSA patients before and after 1 night and 3 months of continuous positive airway pressure treatment.

DETAILED DESCRIPTION:
Measurement of exhaled Nitric Oxide and collection of exhaled breath condensate and peripheral blood. This will be done 2 to 4 times(on admission,the morning after sleep study,immediately after CPAP titration, after CPAP use for 3 months). Each time eNO will be measured first, followed by EBC collection.

For the tests in the morning, patients will be asked to postpone his/her breakfast until after the test which will take less than half an hour.

OSA is defined as patients having a respiratory disturbance index of ≥5/hr.

Measurement of Exhaled Nitric Oxide:

eNO will be measured using a Sievers 280i chemiluminescence analyser (Sievers Instruments, Boulder, CO, USA) sensitive to NO from 1 ppb to 200 ppm and with a resolution of 1 ppb and accuracy of 1 ppb designed for online recording. The eNO measurement will be performed according to ATS standards. Briefly, subjects should remain seated without nose clip during the procedure, with 2-minute rest between eNO measurements. The eNO will be measured online at an expiratory flow rate of 50 ml/sec, a dead space of 10 ml and 2-second plateau duration. Repeated exhalations are performed until three NO plateau values agree at the 10% level or two agree at the 5% level. The mean NO value will then be recorded.

Collection of Exhaled Breath Condensate:

EBC will be collected using the ECoscreen (Jaeger, Germany) according to manufacturer instructions. After rinsing their mouth, the recruited subjects will breathe tidally through a mouthpiece that is connected through a unique one-way valve into a cooled collection tube where vapours, aerosols and moisture in the breath condense along the walls of the tube. The one-way valve is then used as a plunger that collects droplets stuck to the inside wall and holds the sample near the top of the tube. The device inherently prevents salivary contamination as shown by the absence of salivary amylase in EBC. On average, this device will be able to collect 300 microL per minute of EBC for an adult. Each subject will be asked to breathe through the collection kit for 5 minutes, which should be sufficiently long to yield 1 ml of condensate for inflammatory marker analysis. EBC will be stored immediately at -70oC until analysis for inflammatory markers.

Measurement of 8 isoprostane, GRO alpha, MCP1, eotaxin and MDC levels in exhaled breath condensate:

EBC stored at -70oC will be analysed for 8-isoprostane, GROalpha, MCP1, eotaxin and MDC levels concentrations in batches. We will use 96-well polystyrene microplates coated with murine monoclonal antibodies against human 8 isoprostane, GRO alpha, MCP1, eotaxin and MDC levels. The levels of these markers in EBC will be measured in duplicates by sandwich enzyme immunoassay (R & D Systems, Minneapolis, MN, USA) according to instructions provided by the manufacturer.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be recruited upon admission for sleep study under the Division of Respiratory Medicine, Prince of Wales Hospital.
* Patients who are aged 18 to 60 will be recruited.

Exclusion Criteria:

* Known history of respiratory disease that will affect inflammatory markers in EBC like asthma, chronic obstructive pulmonary disease and bronchiectasis.
* Upper or lower respiratory tract infection within 6 weeks from the study.
* Current smokers, or ex-smoker who quitted for less than a year.
* Pregnant subjects.
* Any form of malignancies or serious medical illness that will affect the survival of the subject significantly in 1 year period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Changes in the biomarkers in breath over a period of time in subjects with CPAP and no CPAP treatment for the OSA | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Fanny WS Ko, MBChB, Principal Investigator — CUHK
Locations (1):
- Prince of Wales Hospital, Shatin, N.T., Hong Kong